CLINICAL TRIAL: NCT04181086
Title: Pattern and Management of Intracranial Cavernoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Moataz Elshenawi, assistant lecturer, Assiut University
Other Study IDs: intracranial cavernoma
Record Dates: First submitted 2019-11-03; First posted 2019-11-29 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Management of Intracranial Cavernous Hemangioma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: surgical excision of intracranial cavernoma — microvascular excision of intracranial cavernoma

SUMMARY:
Intracranial cavernous vascular malformations are variously known as cavernous angiomas, cavernous hemangiomas, or, more simply, cavernomas. Cavernomas are congenital low flow vascular lesions. It composed of irregular sinusoidal vascular channels, lacking smooth muscle, and elastic fibers. They lack feeding arteries or draining veins and contain no neural tissue. The first description of an intracranial cavernoma was given by Virchow, in 1863. For over a century, it was considered to be an extremely rare malformation, usually found at autopsy, and exceptionally diagnosed during life. The prevalence of cerebral cavernous malformations (CCM) is estimated to be 0.4-0.9%.

ELIGIBILITY:
Inclusion Criteria:

* All patients presented with intracranial cavernomas (single or multiple, superficial or deep, supratentorial or infratentorial)
* Denovo or recurrent patients.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: all patients with confirmed diagnosis of intracranial cavernoma with MRI and will undergo surgery
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
clinical outcome | one month post operative
  Measured by Modified Rankin Scale Measures the degree of disability or dependence in the daily activities of people who have suffered any cause of neurological disability.
  The scale runs from 0-6, running from perfect health without symptoms to death.
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.

IPD SHARING:
Plan to Share IPD: Undecided